CLINICAL TRIAL: NCT01307826
Title: Comparison of the Effectiveness of Massage Based on the Tensegrity Rule and Classical Massage in Treating Painful Shoulder
Brief Title: Massage in Treating Painful Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: University School of Physical Education in Wroclaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27022011KASS
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2010-09

CONDITIONS: Shoulder Pain Syndrome; Pain; Frozen Shoulder
Keywords: massage; shoulder; pain; range of motion; restricted range of motion
MeSH Terms: conditions — Pain; Bursitis | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- tensegrity massage (Experimental): In this group of patients massage sessions based on the tensegrity method were applied.
  Interventions: Other: massage
- classical massage (Active Comparator): In this group of patients 10 classical massage sessions were applied
  Interventions: Other: massage

INTERVENTIONS:
Other: massage — session - 20 minutes.
  Before the massage, palpable evaluation of the selected anatomical structures was carried out - to determine which tissues have the greatest sensitivity and which motor organs show increased tension (by pressing the attachment). In all the examined patients, pain of the following muscle attachments were shown:
  * latissimus muscle of the back
  * major pectoral muscle
  * supraspinous and infraspinous muscles
  * teres minor muscle
  * serratus anterior muscle
  * deltoid muscle The decision which muscles and fascias have to be massaged was made on the basis of the performed evaluation. In most cases the above mentioned tissues (together with other motor system organs which are structurally linked to it) were massaged to relax them.
  A palpable evaluation of the previously examined points was again performed during the final part, with particular attention paid to painful muscles, in order to analyze the effectiveness of the performed relaxation.
  Arms: tensegrity massage
Other: massage — classical massage (Swedish massage)
  Arms: classical massage

SUMMARY:
The purpose of this study is to compare classical massage and massage based on the tensegrity rule in treating people with painful shoulder.

DETAILED DESCRIPTION:
The joint system of the shoulder girdle is exposed to frequent overloading, which can cause painful shoulder. The therapeutic methods applied in the treatment of painful shoulder syndrome include among others oral pharmacotherapy, joint injections, kinesitherapy, ultrasound, electrotherapy, laser. Manual therapy, chiropractic and surgery could also be used. Attempts have also been made to apply classical massage in treating painful shoulder, although it is not often used due to its low effectiveness.This study compares classical massage and massage based on the tensegrity rule which is not commonly known.

ELIGIBILITY:
Inclusion Criteria:

* painful shoulder syndrome

Exclusion Criteria:

* acute pain
* previous bones fracture
* bone relocations in the area of the shoulder girdle
* neck spondylosis
* hemiparesis
* rheumatoid arthritis
* any neurological symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
mobility measurement | immediately before the first massage session - Test 1, on the day the therapy ended - Test 2 - two weeks after therapy started, and one month after the last massage - Test 3
  To assess massage effectiveness, mobility measurements were conducted in each patient. Both were conducted three times

SECONDARY OUTCOMES:
McGill Pain Questionnaire (SF-MPQ) | immediately before the first massage session - Test 1, on the day the therapy ended - Test 2 - two weeks after therapy started, and one month after the last massage - Test 3
  To assess massage effectiveness, McGill Pain Questionnaire (SF-MPQ) were conducted in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Kassolik, PhD, Study Chair — University School of Physical Education in Wrocław
Locations (1):
- University School of Physical Education in Wrocław, Wroclaw, Wroclaw Destrict, Poland

REFERENCES:
- [Background] Ingber DE. Tensegrity and mechanotransduction. J Bodyw Mov Ther. 2008 Jul;12(3):198-200. doi: 10.1016/j.jbmt.2008.04.038. Epub 2008 Jun 16. PMID 19083675
- [Background] Yamada T, Richiert D, Tumminia SJ, Russell P. The tensegrity model applied to the lens: a hypothesis for the presence of the fiber cell ball and sockets. Med Hypotheses. 2000 Jul;55(1):36-9. doi: 10.1054/mehy.1999.0994. PMID 11021323
- [Background] Chen CS, Ingber DE. Tensegrity and mechanoregulation: from skeleton to cytoskeleton. Osteoarthritis Cartilage. 1999 Jan;7(1):81-94. doi: 10.1053/joca.1998.0164. PMID 10367017
- [Background] Ingber DE. Opposing views on tensegrity as a structural framework for understanding cell mechanics. J Appl Physiol (1985). 2000 Oct;89(4):1663-70. doi: 10.1152/jappl.2000.89.4.1663. No abstract available. PMID 11007610
- [Background] May S, Greasley A, Reeve S, Withers S. Expert therapists use specific clinical reasoning processes in the assessment and management of patients with shoulder pain: a qualitative study. Aust J Physiother. 2008;54(4):261-6. doi: 10.1016/s0004-9514(08)70005-9. PMID 19025506
- [Background] Hand C, Clipsham K, Rees JL, Carr AJ. Long-term outcome of frozen shoulder. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):231-6. doi: 10.1016/j.jse.2007.05.009. Epub 2007 Nov 12. PMID 17993282
- [Background] Bunker TD, Anthony PP. The pathology of frozen shoulder. A Dupuytren-like disease. J Bone Joint Surg Br. 1995 Sep;77(5):677-83. PMID 7559688
- [Background] Stevenson K. Evidence-based review of shoulder pain. Musculoskeletal Care. 2006 Dec;4(4):233-9. doi: 10.1002/msc.96. No abstract available. PMID 17117447
- [Background] Wies J, Treatment of eight patients with frozen shoulder: a case study series. Journal of Bodywork and Movement Therapies 9:58-64, 2004.
- [Background] McMahon PJ, Sallis RE. The painful shoulder. Zeroing in on the most common causes. Postgrad Med. 1999 Dec;106(7):36-8, 41-3, 47-9. doi: 10.3810/pgm.1999.12.800. PMID 10608963
- [Background] Myers TW, Anatomy Trains, Myofascial Meridians for Manual and Movement Therapists. Churchill Livingstone: Edinburgh; 2009.
- [Result] Brox JI. Regional musculoskeletal conditions: shoulder pain. Best Pract Res Clin Rheumatol. 2003 Feb;17(1):33-56. doi: 10.1016/s1521-6942(02)00101-8. PMID 12659820
- [Result] Andrews JR. Diagnosis and treatment of chronic painful shoulder: review of nonsurgical interventions. Arthroscopy. 2005 Mar;21(3):333-47. doi: 10.1016/j.arthro.2004.11.003. PMID 15756189
- [Result] Bunker TD, Frozen shoulder. Current Orthopaedics 12:193-201, 1998.